CLINICAL TRIAL: NCT01113151
Title: Daily Magnesium-supplement With Mablet for Steroid-resistant, Severe Asthmatics
Brief Title: Daily Magnesium-supplement for Severe Asthmatics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Gunnar Kjems APS (Industry); GCP-unit at Aarhus University Hospital, Aarhus, Denmark (Other); Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 9727c
Record Dates: First submitted 2010-04-27; First posted 2010-04-29 (Estimated); Last update posted 2013-09-04 (Estimated); Status verified 2013-09

CONDITIONS: Asthma
Keywords: Steroid-resistant; Severe asthmatics; Annual symptoms; Daily magnesium supplement; ACT (asthma control test)
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Washout (No Intervention)
- Mablet (Active Comparator)
  Interventions: Dietary Supplement: Mablet (Magnesium-supplement)
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Mablet (Magnesium-supplement) — 3 tablets daily for 12 weeks of Mablet (360 mg magnesium hydroxide/ -oxide) Produced by: Gunnar Kjems APS
  Other Names: Mablet
  Arms: Mablet
Other: Placebo — 3 placebo tablets daily for 12 weeks
  Arms: Placebo

SUMMARY:
The present study is part of a project titled 'Magnesium in asthma and chronic obstructive pulmonary disease'. The hypothesis of the main project is that a daily magnesium supplement will benefit patients with asthma and chronic obstructive pulmonary disease.

The aim of this part of the project is to reveal possible beneficial effects of daily magnesium supplement for severe asthmatics, refractory to conventional treatment.

ELIGIBILITY:
Inclusion Criteria:

* severe asthmatics, refractory to conventional treatment, including systemic steroid treatment; symptoms must be annual.

Exclusion Criteria:

* Se-Mg > 2,00 mmol/L,
* smoking cessation less than 1 year prior to study start,
* major changes in eating habits within three months prior to study start and during the study period of approximately one year,
* various conditions (e.g. gastrointestinal disease, kidney disease, pregnancy/lactation) that may affect the study results.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2011-04; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Asthma control test (ACT) | Two years
  Questionnaire providing a level of disease control

SECONDARY OUTCOMES:
EQ-5D | Two years
  Questionnaire providing a degree of quality of life
Spirometry | Two years
  Lung function testing
Reversibility testing | Two years
  Lung function reversibility testing with beta2-agonists
Diary | Two years
  Participants will register asthma symptoms, use of reliever medication and exacerbations
Adverse effects | Two years
Blood- and urine samples | Two years
  Se-magnesium, dU-magnesium, se-creatinin, se-potassium, se-sodium, se-albumine, se-Ca2+, se-phosphate, dU-Ca and dU-creatinine
Endogen NO in expiratory breath and Impulse Oscillometry. | Two years

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Dahl, Professor, Principal Investigator — Dept. of Respiratory Medicine, Aarhus University Hospital, Denmark
Locations (1):
- Research Dept. of Respiratory Medicine, Aarhus University Hospital, Aarhus C, Denmark

REFERENCES:
- [Background] Schlingmann KP, Konrad M, Seyberth HW. Genetics of hereditary disorders of magnesium homeostasis. Pediatr Nephrol. 2004 Jan;19(1):13-25. doi: 10.1007/s00467-003-1293-z. Epub 2003 Nov 22. PMID 14634861
- [Background] Beasley R, Aldington S. Magnesium in the treatment of asthma. Curr Opin Allergy Clin Immunol. 2007 Feb;7(1):107-10. doi: 10.1097/ACI.0b013e328012ce4b. PMID 17218820
- [Background] Emelyanov A, Fedoseev G, Barnes PJ. Reduced intracellular magnesium concentrations in asthmatic patients. Eur Respir J. 1999 Jan;13(1):38-40. doi: 10.1183/09031936.99.13103899. PMID 10836320
- [Background] Dominguez LJ, Barbagallo M, Di Lorenzo G, Drago A, Scola S, Morici G, Caruso C. Bronchial reactivity and intracellular magnesium: a possible mechanism for the bronchodilating effects of magnesium in asthma. Clin Sci (Lond). 1998 Aug;95(2):137-42. PMID 9680494
- [Background] Alamoudi OS. Hypomagnesaemia in chronic, stable asthmatics: prevalence, correlation with severity and hospitalization. Eur Respir J. 2000 Sep;16(3):427-31. doi: 10.1034/j.1399-3003.2000.016003427.x. PMID 11028655
- [Background] Bede O, Suranyi A, Pinter K, Szlavik M, Gyurkovits K. Urinary magnesium excretion in asthmatic children receiving magnesium supplementation: a randomized, placebo-controlled, double-blind study. Magnes Res. 2003 Dec;16(4):262-70. PMID 14979636
- [Background] Aziz HS, Blamoun AI, Shubair MK, Ismail MM, DeBari VA, Khan MA. Serum magnesium levels and acute exacerbation of chronic obstructive pulmonary disease: a retrospective study. Ann Clin Lab Sci. 2005 Autumn;35(4):423-7. PMID 16254259
- [Background] Rowe BH, Camargo CA Jr. The role of magnesium sulfate in the acute and chronic management of asthma. Curr Opin Pulm Med. 2008 Jan;14(1):70-6. doi: 10.1097/MCP.0b013e3282f19867. PMID 18043278
- [Background] Nasulewicz A, Zimowska W, Bayle D, Dzimira S, Madej J, Rayssiguier Y, Opolski A, Mazur A. Changes in gene expression in the lungs of Mg-deficient mice are related to an inflammatory process. Magnes Res. 2004 Dec;17(4):259-63. PMID 15726901
- [Background] Gontijo-Amaral C, Ribeiro MA, Gontijo LS, Condino-Neto A, Ribeiro JD. Oral magnesium supplementation in asthmatic children: a double-blind randomized placebo-controlled trial. Eur J Clin Nutr. 2007 Jan;61(1):54-60. doi: 10.1038/sj.ejcn.1602475. Epub 2006 Jun 21. PMID 16788707
- [Background] Fogarty A, Lewis SA, Scrivener SL, Antoniak M, Pacey S, Pringle M, Britton J. Oral magnesium and vitamin C supplements in asthma: a parallel group randomized placebo-controlled trial. Clin Exp Allergy. 2003 Oct;33(10):1355-9. doi: 10.1046/j.1365-2222.2003.01777.x. PMID 14519140
- [Background] Hill J, Micklewright A, Lewis S, Britton J. Investigation of the effect of short-term change in dietary magnesium intake in asthma. Eur Respir J. 1997 Oct;10(10):2225-9. doi: 10.1183/09031936.97.10102225. PMID 9387944
- [Background] Abreu Gonzalez J, Hernandez Garcia C, Abreu Gonzalez P, Martin Garcia C, Jimenez A. [Effect of intravenous magnesium sulfate on chronic obstructive pulmonary disease exacerbations requiring hospitalization: a randomized placebo-controlled trial]. Arch Bronconeumol. 2006 Aug;42(8):384-7. doi: 10.1016/s1579-2129(06)60551-x. Spanish. PMID 16948990